CLINICAL TRIAL: NCT05087589
Title: Efficacy, Safety and Immunological Evaluation of Tofacitinib in the Treatment of Primary Sjögren's Syndrome:a Prospective Observational Study
Brief Title: Efficacy, Safety and Immunological Evaluation of Tofacitinib in the Treatment of Primary Sjogren's Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210918pss
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-10

CONDITIONS: Primary Sjögren's Syndrome
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tofacitinib (Experimental): Tofacitinib 5mg was taken orally twice a day for 6 months
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib 5mg was taken orally twice a day for 6 months

SUMMARY:
This study aims to explore the clinical and immunological efficacy of tofacitinib on primary Sjögren's Syndrome

DETAILED DESCRIPTION:
The investigators designed a single center, open-label, prospective study. Adults with active primary Sjögren's Syndrome will be enrolled, meeting the American College of Rheumatology(ACR) & European allance of associations for rheumatology(EULAR)(2016) diagnostic criteria . Tofacitinib 5 mg bd was administered for 6 months to explore its efficacy and safety. The improvement of clinical and laboratory indexes was evaluated. Changes of immune cell subsets and cytokines were monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female >18 years of age at screening visits
2. Patients meet the American-European Consensus Group 2002 classification criteria
3. The patient must be informed in writing of the consent to participate in the trial and the patient is expected to be able to comply with the requirements of the study follow-up plan and other protocols.
4. Dosing of antimalarials, prednisone or equivalent, cholinergic stimulants, and topical cyclosporine required to be stable for at least 4 weeks before screening and during study; maximum doses allowed:

   * Hydroxychloroquinone, 400 mg/day;
   * Prednisone, 10 mg/day

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Laboratory abnormality:

   * Hb≤9 g/dl
   * Neutrophil <1.0 x 109/l
   * lymphocyte<0.5 x 109/l
2. Diagnosis of other autoimmune disease, or other sicca syndrome.
3. Use rituximab or other monoclonal antibodies within 6 months.
4. Received high doses of glucocorticoid (>10 mg/d) within 1 month.
5. Serious complications: including heart failure (≥ New York Heart Association (NYHA) class III), renal insufficiency (creatinine clearance ≤ 30 ml/min), liver dysfunction (serum Alanine transaminase (ALT) or aspartate aminotransferase (AST) greater than three times the upper limit of normal, or total bilirubin greater than Normal upper limit)
6. Known allergies, hyperreactivity or intolerance of tofacitinib or its excipients.
7. Have a serious infection needing hospitalization (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, EB virus, tuberculosis infection), or use intravenous antibiotics to treat infection in 2 months before the enrollment.
8. Infection with HIV (HIV antibody positive serology) or hepatitis C (Hep C antibody positive serology). If seropositive, it is recommended to consult a doctor who has expertise in treating HIV or hepatitis C virus infection.
9. Any known history of malignancy in the past 5 years (except for non-melanoma skin cancer, non-melanoma skin cancer or cervical tumor without recurrence within 3 months after surgical cure prior to the first study preparation).
10. Uncontrolled mental or emotional disorders, including a history of drug and alcohol abuse over the past 3 years, may hinder the successful completion of the study.
11. Pregnant, lactating women (WCBP) are reluctant to use medically approved contraceptives during treatment and 12 months after treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-11-20 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Immunological Responses | week 24
  Analysis interleukin 17 (IL-17)-producing helper T (Th17) cells before and during tofacitinib treatment. P values below 0.05 are considered statistically significant in this study.

SECONDARY OUTCOMES:
Improvements in EULAR SS patient-reported index (ESSPRI), other clinical and immunological parameters | week 24
  ESSPRI ranges from 0 to 10. The patient's acceptability/satisfaction of its current state (taking account of his symptoms: dryness, fatigue and pain) should be recorded. For addressing patient-reported outcomes, we define response as an improvement of ESSPRI at least one point or 15% .
Safety and tolerability of tofacitinib as assessed by incidence of adverse events reported and observed | up tp 24 weeks
  we will report frequency of adverse events.Adverse events includes infection, tumor, abnormal neutrophil and lymphocyte count, anemia,drug-induced liver and kidney damage.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Principal Investigator — Peking University Institute of Rheuamotology and Immunology
Locations (1):
- Department of Rheumatology and Immunology, Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu Q, Zeng Y, Xing X, Huang B, Feng R, Wang Y, Wang N, Zhang X, Li Y, Su L, Jacob A, Ambrus JL Jr, Shen L, Suresh L, Yu D, Lin X, He J. Evaluating the therapeutic potential of tofacitinib in Sjogren's disease: a comprehensive clinical and immunological assessment. Rheumatology (Oxford). 2025 Nov 1;64(11):5899-5910. doi: 10.1093/rheumatology/keaf173. PMID 40139690